CLINICAL TRIAL: NCT04517201
Title: Study to Assess Artificial Intelligence-Assisted Insulin Titration System on Inpatients Glucose Control
Brief Title: AI-Assisted Insulin Titration System on Inpatients Glucose Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Hua Bian, Director, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iNCDSS-2
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes
Keywords: iNCDSS; T2D; AI
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI group (Experimental): iGMS+iNCDSS group (Artificial intelligence assisted insulin titration system group)
  Interventions: Drug: iNCDSS based insulin regime
- Control group (Active Comparator): iGMS+routine treatment group (Physicians decided insulin titration group)
  Interventions: Drug: Physician based insulin regime

INTERVENTIONS:
Drug: iNCDSS based insulin regime — Patients of this group will receive the insulin regime set by the AI assisted insulin titration system (iNCDSS).
  Other Names: iGMS + iNCDSS based insulin regime
  Arms: AI group
Drug: Physician based insulin regime — Patients of this group will receive the insulin regime recommended by professional endocrinologists.
  Other Names: iGMS + routine insulin treatment regime
  Arms: Control group

SUMMARY:
This is a multi-center, open-labeled, parallel group, randomized controlled trial to access the effect and safety of the Artificial Intelligence Assisted Insulin Titration System (iNCDSS) in patients with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
As one of the most common treatments for diabetes inpatients, insulin regimens often vary due to different physicians. Since 2016, Zhongshan Hospital has set up the Internet-based glucose management system (iGMS) to monitor plasma glucose of diabetes patients, and further set up an Artificial Intelligence Assisted Insulin Titration System (iNCDSS) to recommend insulin regime in 2019. Previous single-center clinical trial (NCT04053959) have demonstrated the efficacy and safety of iNCDSS in glycemic management in patients with type 2 diabetes.

This multi-center study enrolls 120 patients with Type 2 Diabetes from 20 wards of Zhongshan Hospital who are on treatment with insulin for at least 3 months. They are randomly allocated into 2 groups at a ratio of 1:1 after screening for the inclusion and exclusion criteria. Patients in the Intervention group (AI group) receive insulin regimen set by iNCDSS and patients in Control group receive insulin regimen recommended by endocrinologists.

This study will be conducted in the Department of Endocrinology, Zhongshan Hospital,Fudan University and consist of a 7-day intervention period. Patient allocation will be stratified by HbA1c, BMI and previous total insulin doses. The primary endpoint is the fasting plasma glucose level after the 7-days trial period.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18-99 years old;
* Inpatients who had been diagnosed with type 2 diabetes;
* Subjects who are on treatment with insulin for at least 3 months;
* HbA1c: 7.0%-10.0%.

Exclusion Criteria:

* Patients who were diagnosed with T1D, gestational diabetes or other specific types of diabetes.
* Subjects with acute complications of diabetes such as ketoacidosis or hyperglycemic hyperosmolar state;
* Patients with severe cardiac, hepatic, renal or general diseases;
* Subjects that are, in the judgement of the investigator, unlikely to comply with the protocol.
* Absence of informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Fasting plasma glucose of T2D patients | After 7-day intervention
  Fasting plasma glucose of T2D patients by self-monitoring of bloodglucose (SMBG) in both groups

SECONDARY OUTCOMES:
Well-controlled rate of fasting blood glucose | During 7-day intervention
  The well-controlled rate of blood glucose is defined as proportion of the time of sensor glucose measurements in targeted range
Incidence of hypoglycemia | During 7-day intervention
  The hypoglycemia is defined as blood glucose level less than 3.9mmol/L.
Total insulin dose | During 7-day intervention
  The total insulin dose is defined as daily insulin dose.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Bian, Principal Investigator — Shanghai Zhongshan Hospital
Locations (2):
- China (2):
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu Y, Wang L, He J, Bi Y, Li M, Wang T, Wang L, Jiang Y, Dai M, Lu J, Xu M, Li Y, Hu N, Li J, Mi S, Chen CS, Li G, Mu Y, Zhao J, Kong L, Chen J, Lai S, Wang W, Zhao W, Ning G; 2010 China Noncommunicable Disease Surveillance Group. Prevalence and control of diabetes in Chinese adults. JAMA. 2013 Sep 4;310(9):948-59. doi: 10.1001/jama.2013.168118. PMID 24002281
- [Background] Wang T, Xu Y, Xu M, Wang W, Bi Y, Lu J, Dai M, Zhang D, Ding L, Xu B, Sun J, Zhao W, Jiang Y, Wang L, Li Y, Zhang M, Lai S, Wang L, Ning G. Awareness, treatment and control of cardiometabolic disorders in Chinese adults with diabetes: a national representative population study. Cardiovasc Diabetol. 2015 Feb 26;14:28. doi: 10.1186/s12933-015-0191-6. PMID 25848699
- [Background] Fox CS, Golden SH, Anderson C, Bray GA, Burke LE, de Boer IH, Deedwania P, Eckel RH, Ershow AG, Fradkin J, Inzucchi SE, Kosiborod M, Nelson RG, Patel MJ, Pignone M, Quinn L, Schauer PR, Selvin E, Vafiadis DK; American Heart Association Diabetes Committee of the Council on Lifestyle and Cardiometabolic Health, Council on Clinical Cardiology, Council on Cardiovascular and Stroke Nursing, Council on Cardiovascular Surgery and Anesthesia, Council on Quality of Care and Outcomes Research, and the American Diabetes Association. Update on Prevention of Cardiovascular Disease in Adults With Type 2 Diabetes Mellitus in Light of Recent Evidence: A Scientific Statement From the American Heart Association and the American Diabetes Association. Circulation. 2015 Aug 25;132(8):691-718. doi: 10.1161/CIR.0000000000000230. Epub 2015 Aug 5. PMID 26246173
- [Background] Rawshani A, Rawshani A, Gudbjornsdottir S. Mortality and Cardiovascular Disease in Type 1 and Type 2 Diabetes. N Engl J Med. 2017 Jul 20;377(3):300-301. doi: 10.1056/NEJMc1706292. No abstract available. PMID 28723317
- [Background] Contreras I, Vehi J. Artificial Intelligence for Diabetes Management and Decision Support: Literature Review. J Med Internet Res. 2018 May 30;20(5):e10775. doi: 10.2196/10775. PMID 29848472